CLINICAL TRIAL: NCT05609513
Title: PULESA Uganda: Strengthening the Blood Pressure Care and Treatment Cascade for Ugandans Living With HIV-ImpLEmentation Strategies to SAve Lives
Brief Title: Integration of Hypertension Management in HIV Care in Uganda
Acronym: PULESAUganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Infectious Diseases Research Collaboration, Uganda (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Mak-SOMREC-2022-420; 4UH3HL154501-03 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2024-06

CONDITIONS: HIV/AIDS; Hypertension
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypertension

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster randomized trial. Sixteen clinics will be randomized to the order in which they will begin intervention, with two clinics initiating the intervention every 2 months after a 2-month run-in period. Sites will be additionally randomized to receive the HTN-BASIC package only or the enhanced HTN-PLUS intervention. We will collect clinic data during the control period, run-in period and the intervention phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8 HIV clinics randomized to HTN BASIC (Experimental): The HTN-BASIC intervention will consist of providing consistent access to diagnostic equipment and evidence-based antihypertensive drugs at no cost to the hypertensive patients. Access to a consistent supply of three anti-hypertensive drugs (amlodipine 5, 10mg; valsartan 80, 160mg; and hydrochlorothiazide 12.5, 25mg) will be supplied to each clinic in the trial.
  Interventions: Other: HTN-BASIC
- 8 HIV clinics randomized to HTN PLUS (Experimental): In addition to receiving all the components of HTN-BASIC, HTN-PLUS sites will receive an enhanced, more human-resource intensive package of interventions that have been developed in consultation with key stakeholders during our human-centered design phase. The intervention components will include four broad categories- (1) hypertension training, (2) differentiated service delivery and (3) remote patient monitoring for hypertension and (4) Performance Improvement Program. Uptake of all components will be assessed on a monthly basis during the intervention period. These interventions will by nature cost more, and so cost data will be rigorously collected as well.
  Interventions: Other: HTN-PLUS
- Control Period for all 16 clinics (No Intervention): Outcome data will be collected during the control period prior to intervention roll-out in all 16 clinics.

INTERVENTIONS:
Other: HTN-BASIC — The HTN-BASIC intervention will consist of providing consistent access to diagnostic equipment and evidence-based antihypertensive drugs at no cost to the hypertensive patients. Access to a consistent supply of three anti-hypertensive drugs (amlodipine 5, 10mg; valsartan 80, 160mg; and hydrochlorothiazide 12.5, 25mg) will be supplied to each clinic in the trial.
  Arms: 8 HIV clinics randomized to HTN BASIC
Other: HTN-PLUS — In addition to receiving all the components of HTN-BASIC, HTN-PLUS sites will receive an enhanced, more human-resource intensive package of interventions that have been developed in consultation with key stakeholders during our human-centered design phase. The intervention components will include four broad categories- (1) hypertension training, (2) differentiated service delivery and (3) remote patient monitoring for hypertension and (4) Performance Improvement Program. Uptake of all components will be assessed on a monthly basis during the intervention period. These interventions will by nature cost more, and so cost data will be rigorously collected as well.
  Arms: 8 HIV clinics randomized to HTN PLUS

SUMMARY:
Effective, cost-effective, scalable, sustainable, and equitable implementation strategies to improve care for people living with HIV and co-morbid hypertension in sub-Saharan Africa are urgently needed. Our study will compare the effectiveness, scalability, and cost-effectiveness of a lower-resource intensive vs. a higher resource intensive strategy to integrate hypertension care into HIV clinics in Uganda.

DETAILED DESCRIPTION:
Chronic HIV infection is a well-established risk factor for cardiovascular disease (CVD). In sub-Saharan Africa(SSA)-a region that may account for half of the global burden of CVD attributable to HIV-hypertension is the most important driver of CVD risk. Profound barriers to effective hypertension management exist, including limited knowledge, inconsistent BP measurement, and poor access to medications. HIV care innovations such as access to no-cost antiretroviral therapy, differentiated service delivery and use of PLHIV peers in care models may improve care of comorbid conditions such as hypertension. The overarching goal of PULESA-UGANDA study is to improve the BP treatment cascade for people living with HIV (PLHIV) in urban and peri-urban Uganda in a scalable and sustainable manner. This hybrid IS Type 3 study proposes to first explore current practice, routines, barriers, and facilitators of evidence-based BP care in HIV clinical settings in Kampala and Wakiso districts (Aim 1). Then, using a human-centered design approach, a design team of key stakeholders will use data from the formative assessment to develop a multi-component implementation strategy (HTN-PLUS) to improve uptake and adherence to evidence-based BP treatments, contextually adapted to these Ugandan HIV clinics (Sub-aim 1.1). The design team will adapt differentiated service delivery models, use of hypertensive PLHIV peer champions, and methods of BP monitoring that address specific barriers and facilitators of BP care. In a stepped-wedge cluster randomized trial of 16 clinics from Kampala and Wakiso, the investigators will determine the effectiveness of implementation strategies to improve BP cascade metrics (Aim 2). Clinics will be randomized to receive free and consistent access to diagnostic equipment and evidence-based antihypertensive drugs (HTN-BASIC) with and without the multi-component implementation strategy developed in sub-aim 1 (HTN-PLUS). The primary effectiveness outcome will be % of patients with hypertension diagnosis who are controlled (<140mmHg systolic). The investigators hypothesize that the HTN-BASIC intervention will increase control from 25% at baseline to 35%, and that HTN-PLUS will further increase control to 40%. The investigators will conduct an extensive mixed-methods process evaluation. The investigators will assess scalability as our main implementation outcome, and will also assess acceptability, adoption, and implementation climate. Finally, the investigators will evaluate the economic and financial sustainability of the integrated care strategies in a cost-effectiveness analysis from a societal perspective that will include household out-of-pocket expenditures. The primary outcome of this aim will be incremental cost per BP controlled patient. This study will provide much needed evidence to SSA government stakeholders for a strategy to preserve the health gains of HIV treatment by preventing death and disability from CVD.

Importantly, it will offer economic evidence of the scalability, sustainability, and equity of a model of HIV hypertension integration management.

ELIGIBILITY:
Inclusion Criteria:

1) All patients over 18 years of age receiving care at participating HIV clinics will contribute data for the effectiveness outcomes

Exclusion Criteria:

1) Patients who are not diagnosed with HIV receiving care at participating HIV clinics and are under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87421 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Population blood pressure control | Year 3-5
  Proportion (%) of the entire clinic population in care (>18 years old) with a documented BP <140mmhg systolic AND <90mmhg diastolic.
Hypertension patient BP control | Year 3-5
  Proportion (%) of patients with hypertension with a documented BP <140mmhg systolic AND <90mmhg diastolic. <140/90 mmHg

SECONDARY OUTCOMES:
cost-effectiveness | Year 3-5
  Incremental cost per BP-controlled patient

CONTACTS AND LOCATIONS:
Overall Officials: Fred C. Semitala, MBChB, MMED, Principal Investigator — INFECTIOUS DISEASES RESEARCH COLLABORATION
Locations (16):
- Uganda (16):
  - Butabika, Kampala
  - Kawala, Kampala
  - Kisenyi, Kampala
  - Kitebi, Kampala
  - Komamboga, Kampala
  - Mengo Hospital, Kampala
  - Naguru, Kampala
  - Nsambya, Kampala
  - Bweyogerere, Wakiso
  - Entebbe RRH, Wakiso
  - Kakiri, Wakiso
  - Kawanda, Wakiso
  - Nakawuka HCIII, Wakiso
  - Nsangi HCIII, Wakiso
  - Nurture Africa, Wakiso
  - Saidina, Wakiso

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be made available upon request.

REFERENCES:
- [Derived] Longenecker CT, Kiggundu JB, Ayebare F, Muddu M, Kayima J, Mutungi G, Ssinabulya I, Schwartz JI, Spiegelman D, Tong G, Nugent R, Aifah A, Kagoya F, Cameron DB, Hutchinson B, Kamya MR, Katahoire AR, Semitala FC. Implementation strategies to integrate HIV and hypertension care in Kampala and Wakiso districts, Uganda: study protocol for a stepped wedge cluster randomized trial (PULESA-Uganda). BMC Health Serv Res. 2025 Aug 11;25(1):1060. doi: 10.1186/s12913-025-13281-9. PMID 40790739
- [Derived] Kiggundu JB, Semitala FC, Lipoto CF, Giibwa L, Twine R, Mwaka S, Ayebare F, Kiwala C, Magambo EN, Mutungi G, Ssinabulya I, Spiegelman D, Kayima J, Muddu M, Schwartz JI, Katahoire AR, Longenecker CT. Early findings from the integration of hypertension care into differentiated service delivery models for HIV in Uganda: a mixed-method study. J Int AIDS Soc. 2025 Jul;28 Suppl 3(Suppl 3):e26499. doi: 10.1002/jia2.26499. PMID 40622382